CLINICAL TRIAL: NCT05735249
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Two-Part (SAD and MAD) Study to Assess the Safety, Tolerability, and Pharmacokinetics of ARN-75039 When Administered By The Orally Route in Healthy Adult Subjects
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of Oral ARN-75039 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arisan Therapeutics, Inc. (Industry)
Collaborators: The Defense Threat Reduction Agency (DTRA) (Unknown); United States Department of Defense (U.S. Federal Agency); Battelle Memorial Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARN-75039-101
Record Dates: First submitted 2023-01-27; First posted 2023-02-21 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Lassa Virus Infection
Keywords: Lassa virus; Lassa fever; Arenavirus; Hemorrhagic fever
MeSH Terms: conditions — Lassa Fever; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability, and PK of escalating single and multiple doses of ARN-75039 when administered by the oral route in healthy adult subjects. Up to 5 single ascending dose (SAD) cohorts and up to 3 multiple ascending dose (MAD) cohorts, with approximately 8 subjects per cohort, will be enrolled to receive study drug or placebo. Within each cohort, the first 2 subjects will be randomized 1:1 to receive ARN-75039 capsules or placebo. After a review of the first 3 days of blinded safety for these subjects by the Medical Monitor, an additional 6 subjects will be randomized in a 5:1 (active: placebo) ratio. Each subsequent dose escalation will be based on safety data review of the current dose level.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Central, computer-generated randomization scheme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARN-75039 (Experimental): Escalating single or multiple doses of ARN-75039 oral capsules
  Interventions: Drug: ARN-75039 oral capsules
- Placebo (Placebo Comparator): Matching placebo capsules in a same SAD and MAD dosing regimen as ARN-75039
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARN-75039 oral capsules — SAD: Up to 5 single escalating doses MAD: Up to 3 escalating doses Food-effect: Selected single dose
  Other Names: SAD: Cohorts 1 through 5 MAD: Cohorts 7 through 9
  Arms: ARN-75039
Drug: Placebo — Given at frequency and amounts matching ARN- 75039 dosing regimen
  Other Names: Matching placebo oral capsules (Cohorts 1 through 9)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability, and pharmacokinetics (PK) of escalating single ascending dose (SAD) and multiple ascending doses (MAD) of ARN-75039 when administered by the oral route in healthy adult subjects. The SAD portion of the study will enroll approximately 40 subjects for a total duration of 6 weeks. A cohort of 8 subjects in the SAD portion of the study will be selected to assess food effect (including relative bioavailability). The MAD portion of the study will enroll approximately 24 subjects for a total duration of 10 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind study of ARN-75039 or placebo given as single and multiple escalating doses in normal healthy subjects. The study will be conducted in three parts: Part 1 will be a Single Ascending Dose (SAD) study enrolling approximately 40 subjects for a total duration of 6 weeks. Part 2 will be a Multiple Ascending Dose (MAD) study enrolling approximately 24 subjects for a total duration of 10 weeks, and part 3 will be a selected SAD cohort in a fasted state to evaluate the effect of food on the bioavailability of ARN-75039, enrolling approximately 8 subjects from a selected SAD cohort for a duration of 6 weeks. The dose escalation will be performed in a step-wise manner. Dose escalation stopping rules will be used to determine whether or not investigation of a higher dose level will proceed per protocol. Safety and tolerability will be assessed by periodic measurement of vital signs, physical examinations, electrocardiograms, blood laboratory analyses and occurrence of adverse events (AE). PK blood samples will be collected at pre-specified time points for noncompartmental data analysis. The PK parameters include but are not limited to: Cmax, Tmax, AUC, CL, and t½. For determination of the food effect, for selected PK parameters (e.g., Cmax, AUC0-τ, and AUC0-∞), comparisons between the fed and fasted conditions will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, age 18 to 55 years, inclusive, at Screening.
2. Body mass index (BMI) between 18.5 and 35 kg/m2, inclusive, at Screening.
3. In good general health, determined by no clinically significant findings in the opinion of the Investigator from medical history, physical examination, 12-lead electrocardiogram (ECG), clinical laboratory findings, and vital signs at Screening and Day -1 or 1.
4. Hemoglobin, hematocrit, white blood cell count, absolute neutrophil count, and platelet count results within the laboratory reference range at Screening; subjects with Gilbert's disease with associated abnormalities of liver function tests are eligible for enrollment. Tests may be repeated at the discretion of the Investigator to confirm abnormalities.
5. Estimated glomerular filtration rate (eGFR) based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation of ≥ 80 mL/min/1.73m2 at Screening
6. Females of childbearing potential must practice effective contraception per national regulatory guidelines for clinical trials from Screening, throughout the study and for 28 days after the EOS visit.
7. Females of childbearing potential must have a negative pregnancy test at Screening and within 24 hours prior to dosing of study drug; for post-menopausal subjects, a blood sample will also be tested for follicle stimulating hormone (FSH) to confirm post-menopausal status (as verified by an FSH of ≥40). Surgically sterile females are eligible; however, proof via medical records will be required.
8. Males must agree to not donate sperm and/or to use condoms during sexual intercourse from the time of the first study drug administration and for 90 days following the last dose of study drug, and females must agree not to donate eggs from the time of the first study drug administration and for 60 days following the last dose of study drug.
9. Must be willing and able to comply with measures to avoid photosensitivity reactions (i.e., avoidance of outdoor sun exposure and tanning; consistent use of long sleeve shirts, long pants, hats, and sunglasses; consistent use of SPF 75 or greater sunscreen when outdoors) from Day 1 through Day 8 in Part 1 and through Day 29 in Part 2.
10. Able to provide informed consent.
11. Willing and able to comply with this protocol and be available for the entire duration of the study.

Exclusion Criteria:

1. Any clinically significant underlying illness in the opinion of the Investigator.
2. Poor venous access.
3. Inability to ingest all capsules of a multi-capsule dose within 5 minutes of ingestion of the first capsule.
4. Prior exposure to ARN-75039.
5. Positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) at Screening; subjects with adequately treated HCV are eligible for enrollment.
6. Positive test for SARS-CoV-2 infection on Day -1.
7. Consumption of Seville oranges, grapefruit or grapefruit juice within 72 hours prior to Day 1 or during the study.
8. History of drug or alcohol abuse within 1 year of Screening in the opinion of the investigator, or a positive test for drugs of abuse or alcohol at Screening or Day -1.
9. Use of any prescription or over-the-counter (OTC) medications, including food supplements, vitamins, herbal medications (e.g., St. John's wort), and cannabis, with the exception of contraceptive medications and as needed (prn) acetaminophen or paracetamol (not exceeding 2 grams/day) within 7 days prior to study drug administration and through the EOS visit.
10. History of malignancy, except adequately treated basal cell carcinoma or in situ carcinoma of the uterine cervix.
11. Smoking greater than 20 cigarettes, cigars, cigarillos or E-cigarettes per week in the 3 months prior to study drug administration or during the study.
12. Any female who is pregnant or breastfeeding, or any female who is planning to become pregnant during the study and safety follow-up period.
13. Any reason or condition that, in the investigator's opinion, may compromise study participation, present a safety risk to the subject, or may confound the interpretation of the study results.
14. A QT duration corrected for heart rate by Fridericia's formula (QTcF) > 450 millisecond (msec) based on either single or averaged QTcF values of triplicate ECGs obtained over a 3-minute interval (at Screening).
15. Blood product donation within 30 days before Screening.
16. Unwilling to consume a high-fat breakfast on study drug administration days.
17. Currently enrolled in another investigational device or drug study, or less than 30 days or 5 half-lives of the prior investigational agent (whichever is longer) or plans to enroll in another investigational device or drug study during the course of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
The type and frequency of treatment-emergent adverse events (TEAEs) | Day 1 through 14 days post dose for SAD cohorts, and 28 days post last study dose for MAD cohorts.
  Incidence of AEs and SAEs

SECONDARY OUTCOMES:
Determination of the recommended phase 2 dose (RP2D) | Day 1 through 14 days post dose for SAD cohorts and 28 days post last study dose for MAD cohorts.
  Maximum tolerated dose
Determine Maximum Plasma concentrations of ARN-75039 | Day 1 through Day 8 post dose for SAD and FE cohorts, and 28 days post last study dose for MAD cohorts.
  PK of ARN-75039 in health subjects as assessed by maximum plasma concentration (Cmax) towards determination of the optimal PK dose
Determination of time to maximum concentration (Tmax) | Day 1 through Day 8 post dose for SAD and FE cohorts, and 28 days post last study dose for MAD cohorts.
  PK of ARN-75039 in healthy subjects as assessed by time to maximum concentration (Tmax) towards determination of the optimal PK dose
Determination of plasma exposure (AUC0-t, AUC0-inf) | Day 1 through Day 8 post dose for SAD and FE cohorts, and 28 days post last study dose for MAD cohorts.
  PK of ARN-75039 in healthy subjects as assessed by plasma exposure (AUC0-t, AUC0-inf) determination of the optimal PK dose
Determination of terminal half life | Day 1 through Day 8 post dose for SAD and FE cohorts, and 28 days post last study dose for MAD cohorts.
  PK of ARN-75039 in healthy subjects as assessed by terminal elimination half life (t1/2) determination of the optimal PK dose

CONTACTS AND LOCATIONS:
Overall Officials: Ken McCormack, PhD, Study Chair — Arisan Therapeutics, Inc.
Locations (1):
- Spaulding Clinical, LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No